CLINICAL TRIAL: NCT02753088
Title: International, Multicentre, Double-blind, Placebo-controlled, Comparative, Randomized Study to Compare Efficacy and Safety of the Generic Drug BCD-063 (CJSC "BIOCAD", Russia) and Copaxone®-Teva ("Teva Pharmaceutical Industries Limited", Israel) in Patients With Relapsing-remitting Multiple Sclerosis
Brief Title: Efficacy and Safety of BCD-063 and Copaxone-Teva in Patients With Relapsing-Remitting Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BCD-063-1
Record Dates: First submitted 2016-04-19; First posted 2016-04-27 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Relapsing-remitting Multiple Sclerosis
Keywords: Equivalence; BCD-063; Copaxone-Teva
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Glatiramer Acetate; Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BCD-063 (glatiramer acetate) (Experimental): Subcutaneous injection of glatiramer acetate BCD-063 subcutaneously every day
  Interventions: Drug: BCD-063
- Copaxone-Teva (glatiramer acetate) (Active Comparator): Subcutaneous injection of glatiramer acetate Copaxone-Teva subcutaneously every day
  Interventions: Drug: Copaxone-Teva
- Placebo (Placebo Comparator): Subcutaneous injection of mannitol 40 mg, water for injections till 1 ml, every day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BCD-063
  Other Names: glatiramer acetate
  Arms: BCD-063 (glatiramer acetate)
Drug: Copaxone-Teva
  Other Names: glatiramer acetate
  Arms: Copaxone-Teva (glatiramer acetate)
Drug: Placebo
  Other Names: mannitol
  Arms: Placebo

SUMMARY:
The objective of the clinical study of the medicinal product for medical use: to compare efficacy and safety of the generic drug BCD-063 and Copaxone®-Teva in patients with relapsing-remitting multiple sclerosis.

Period of the clinical study of the medicinal product for medical use: from June 10, 2013 to March 23, 2016.

Number of patients, involved into the study of the medicinal product for medical use: 158 patients.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed multiple sclerosis (MS, McDonald criteria 2005);
* Disease more, than 1 year prior to inclusion;
* Presence of 1 relapse previously OR at least 1 Gd+ lesion in T1 regimen;
* EDSS 0-5,5;
* Absence of exacerbations for 4 weeks prior to inclusion;
* Readiness of patients (both genders) to use reliable methods of contraception (at least 1 barrier method in combination with: spermicides, intrauterine device/oral contraceptives)

Exclusion Criteria:

* Secondary progressive and primary progressive forms of multiple sclerosis;
* Other diseases (except multiple sclerosis), which may affect the assessment of the severity of the symptoms of the underlying disease: mask, amplify, modify the symptoms of the underlying disease or cause the clinical manifestations and changes in the data of laboratory and instrumental methods of investigation similar to those of multiple sclerosis;
* Any acute or chronic infection in the acute stage;
* Verified HIV, hepatitis B and C, syphilis;
* Metabolic abnormalities (disorders), which manifest themselves as:

  1. raising the general level of creatinine is more than 2 times over the upper limit of the normal range;
  2. increase in transaminases (ALT, AST) or gamma-glutamyltransferase more than 2.5 times over the upper limit of the normal range;
* Violation of bone marrow function as reducing the total number of leukocytes <3000 /mcl, or a platelet count <125000 /mcl, hemoglobin concentration reduction, or <100 g / l;
* EDSS> 5,5 points;
* Liver disease in the stage of decompensation;
* Congestive heart failure, or not controlled by a drug therapy angina or arrhythmia;
* Pregnancy, breast-feeding or planned pregnancy during the study period;
* Use of any time prior to study any drug for modifying multiple sclerosis: interferon beta-1a, interferon beta-1b, glatiramer acetate, azathioprine, corticosteroids and immunomodulators (except for treating exacerbations corticosteroids), drugs and monoclonal antibodies, cytotoxic and / or immunosuppressive drugs, including, but not limited to drugs: mitoxantrone, cyclophosphamide, cyclosporine, fingolimod, cladribine; or total lymphoid irradiation system;
* System (IV, oral) corticosteroids within 30 days prior to the screening visit;
* Intolerance or allergy to glatiramer acetate, mannitol or other components of the BCD-063 preparations or Copaxone®-Teva;
* History of drug addiction, alcoholism and abuse of drugs;
* Contraindications to MRI (gadolinium allergic to or intolerant of closed spaces, any renal failure, which may interfere with the removal of gadolinium - an acute or chronic renal failure);
* Any malignancies, including in anamnesis;
* Vaccination within 4 weeks prior to study entry (prior to randomization);
* Participation in any other clinical trial within 30 days prior to screening or simultaneous participation in other clinical trials;
* Previous participation in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2013-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Cumulative Unique Activity lesions | 48 weeks
  Cumulative Unique Activity (CUA) detected by MRI

SECONDARY OUTCOMES:
Annual relapse rate | 48 weeks
  Relapse per patient per year
Proportion of patients without relapses | 48 weeks
  Proportion of patients without confirming relapses with magnetic resonance imaging (MRI)
Changing in volume of hypointense T1 lesions | 48 weeks
Changing in volume of T2 lesions | 48 weeks
Amount of new or extended lesions in T2 regimen | 48 weeks
Patients proportion without lesions | 48 weeks
T1 lesions amount | 48 weeks
Expanded Disability Status Scale dynamics | Week 24, Week 48
  Expanded Disability Status Scale (EDSS) scale count at 24th and 48th week, comparing count at week 24 to week 48 for each group
Progression on Multiple Sclerosis Functional Composite scale comparing to the baseline | 48 weeks
Risk of relapse | 48 weeks
  Relative Risk Ratio for relapse in each group
Time till the first relapse | 48 weeks
Multiple Sclerosis Functional Composite scale dynamics | 24, 48 weeks
  Multiple Sclerosis Functional Composite (MSFC) scale count at 24th and 48th week, comparing count at week 24 to week 48 for each group

CONTACTS AND LOCATIONS:
Overall Officials: Roman A. Ivanov, PhD, Study Director — Biocad